CLINICAL TRIAL: NCT05903755
Title: To Understand the Effect of Speed Dependent Treadmill Training on Dual Task Performance in Patient With Parkinson's Disease.
Brief Title: the Effect of Speed Dependent Treadmill Training on Dual Task Performance in Patient With Parkinson's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/23/0223
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: Treadmill training; Dual-task performance; Parkinson disease; Physiotherapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- speed dependent treadmill training on moderate speed (Experimental): speed dependent treadmill training on moderate speed along with strengthening, stretching and range of motion exercises.
  Interventions: Device: speed dependent treadmill training on moderate speed
- speed dependent treadmill training on slow speed (Active Comparator): Speed dependent treadmill training on slow speed along with physiotherapy.
  Interventions: Device: speed dependent treadmill training on slow speed

INTERVENTIONS:
Device: speed dependent treadmill training on moderate speed — Experimental group will receive 14 session of speed dependent treadmill training on moderate speed (3 to 6) for 25 minutes along with strengthening, stretching and range of motion exercises.
  Arms: speed dependent treadmill training on moderate speed
Device: speed dependent treadmill training on slow speed — Control group will receive 14 session of speed dependent treadmill training on slow speed (1 to 2) for 25 min along with physiotherapy.
  Arms: speed dependent treadmill training on slow speed

SUMMARY:
The aim of this randomized clinical trail is to identify the impact of treadmill training on walking while doing dual task in patients with Parkinson's disease. By improving walking speed, bradykinesia would be reduced in Parkinson's patients. So, the findings of this study can help in formulation of future guidelines for management of Parkinson's that will help the clinicians to treat such patients in more efficient way.

DETAILED DESCRIPTION:
A RCT that investigated the effect of Treadmill training and physiotherapy in patient with PD using dual tasking as outcome measure.105 Parkinson's disease (PD) patients; these are the subject who received treadmill training and physiotherapy for 14 days. Both intervention helps the patients to enhance the dual task gait velocity.

A study is to identify the effects of incremental speed-dependent treadmill training on postural instability and fear of falling in Parkinson's disease to observe the postural stability by incremental speed dependent treadmill training. 54 patient of Parkinson's disease (PD) was randomly allocated in to experimental and control group. 8-week training program was conducted including stretching, Range of motion exercises (ROM), and treadmill training. Walking distance of the training group was gradually increased after 16 training sessions. The training group's scores on the Berg Balance Test, Dynamic Gait Index, and Falls Efficacy Scale dramatically improved after the training program. While the control group, shows no significant improvement in outcome measurements. Specific exercise regimens, such as incremental speed-dependent treadmill training, may increase mobility and minimize fear of fall in-patient with Parkinson's disease.

GAP:The study's relatively small sample size is one of its limitations. There is least work done on speed dependent treadmill training and its effect on dual task performance in-patient with Parkinson's disease. More research is require, to compare various treatment options with incremental speed-dependent treadmill training for Parkinson's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk on treadmill for 20 min
* Cognitively able to perform required task
* Hoehn and yarn disease stage between I to III.

Exclusion Criteria:

* Gait impairment
* Cardiac impairment
* Dementia
* History of fall
* Severe Freezing episodes
* Camptocormia (axial deformity)
* Central or peripheral paresis
* Score less than 20 in mini mental scale.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson disease rating scale (UPDRS-III) | 1 day
  UPDRS-III is a "Gold standered" for Parkinson disease. It completely access the body function, activities and participation of Parkinson's patient. It consist of 6 session. We will only use Scale's motor component, which consist of 14 item. Each sign and symptom is rated on a 5-point scale (ranging from 0 to 4) higher score represent severe impairment. Highest point represent total or maximal disability.

SECONDARY OUTCOMES:
dual task gait speed test | 1 day
  This test use to access the dual-task gait speed. the gait speed will be measured in single task first, and then in dual task before and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, Phd, Principal Investigator — Riphah International University
Locations (1):
- General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baek CY, Chang WN, Park BY, Lee KB, Kang KY, Choi MR. Effects of Dual-Task Gait Treadmill Training on Gait Ability, Dual-Task Interference, and Fall Efficacy in People With Stroke: A Randomized Controlled Trial. Phys Ther. 2021 Jun 1;101(6):pzab067. doi: 10.1093/ptj/pzab067. PMID 33611557
- [Background] Gassner H, Trutt E, Seifferth S, Friedrich J, Zucker D, Salhani Z, Adler W, Winkler J, Jost WH. Treadmill training and physiotherapy similarly improve dual task gait performance: a randomized-controlled trial in Parkinson's disease. J Neural Transm (Vienna). 2022 Sep;129(9):1189-1200. doi: 10.1007/s00702-022-02514-4. Epub 2022 Jun 13. PMID 35697942
- [Background] Cakit BD, Saracoglu M, Genc H, Erdem HR, Inan L. The effects of incremental speed-dependent treadmill training on postural instability and fear of falling in Parkinson's disease. Clin Rehabil. 2007 Aug;21(8):698-705. doi: 10.1177/0269215507077269. PMID 17846069
- [Background] Verstraeten A, Theuns J, Van Broeckhoven C. Progress in unraveling the genetic etiology of Parkinson disease in a genomic era. Trends Genet. 2015 Mar;31(3):140-9. doi: 10.1016/j.tig.2015.01.004. Epub 2015 Feb 20. PMID 25703649
- [Background] Rochester L, Nieuwboer A, Baker K, Hetherington V, Willems AM, Kwakkel G, Van Wegen E, Lim I, Jones D. Walking speed during single and dual tasks in Parkinson's disease: which characteristics are important? Mov Disord. 2008 Dec 15;23(16):2312-8. doi: 10.1002/mds.22219. PMID 18816800
- [Background] Plotnik M, Giladi N, Dagan Y, Hausdorff JM. Postural instability and fall risk in Parkinson's disease: impaired dual tasking, pacing, and bilateral coordination of gait during the "ON" medication state. Exp Brain Res. 2011 May;210(3-4):529-38. doi: 10.1007/s00221-011-2551-0. Epub 2011 Jan 30. PMID 21279632
- [Background] Dai S, Piscicelli C, Clarac E, Baciu M, Hommel M, Perennou D. Balance, Lateropulsion, and Gait Disorders in Subacute Stroke. Neurology. 2021 Apr 27;96(17):e2147-e2159. doi: 10.1212/WNL.0000000000011152. Epub 2020 Nov 11. PMID 33177223
- [Background] Cho HY, Kim JS, Lee GC. Effects of motor imagery training on balance and gait abilities in post-stroke patients: a randomized controlled trial. Clin Rehabil. 2013 Aug;27(8):675-80. doi: 10.1177/0269215512464702. Epub 2012 Nov 5. PMID 23129815
- [Background] Mehrholz J, Kugler J, Storch A, Pohl M, Elsner B, Hirsch K. Treadmill training for patients with Parkinson's disease. Cochrane Database Syst Rev. 2015 Aug 22;(8):CD007830. doi: 10.1002/14651858.CD007830.pub3. PMID 26297797
- [Background] Bishnoi A, Lee R, Hu Y, Mahoney JR, Hernandez ME. Effect of Treadmill Training Interventions on Spatiotemporal Gait Parameters in Older Adults with Neurological Disorders: Systematic Review and Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2022 Feb 28;19(5):2824. doi: 10.3390/ijerph19052824. PMID 35270516
- [Background] Mehrholz J, Thomas S, Elsner B. Treadmill training and body weight support for walking after stroke. Cochrane Database Syst Rev. 2017 Aug 17;8(8):CD002840. doi: 10.1002/14651858.CD002840.pub4. PMID 28815562
- [Background] Alghadir AH, Al-Eisa ES, Anwer S, Sarkar B. Reliability, validity, and responsiveness of three scales for measuring balance in patients with chronic stroke. BMC Neurol. 2018 Sep 13;18(1):141. doi: 10.1186/s12883-018-1146-9. PMID 30213258
- [Background] Pohl M, Rockstroh G, Ruckriem S, Mrass G, Mehrholz J. Immediate effects of speed-dependent treadmill training on gait parameters in early Parkinson's disease. Arch Phys Med Rehabil. 2003 Dec;84(12):1760-6. doi: 10.1016/s0003-9993(03)00433-7. PMID 14669180
- [Background] Aprile I, Conte C, Cruciani A, Pecchioli C, Castelli L, Insalaco S, Germanotta M, Iacovelli C. Efficacy of Robot-Assisted Gait Training Combined with Robotic Balance Training in Subacute Stroke Patients: A Randomized Clinical Trial. J Clin Med. 2022 Aug 31;11(17):5162. doi: 10.3390/jcm11175162. PMID 36079092
- [Background] Hulzinga F, Seuthe J, D'Cruz N, Ginis P, Nieuwboer A, Schlenstedt C. Split-Belt Treadmill Training to Improve Gait Adaptation in Parkinson's Disease. Mov Disord. 2023 Jan;38(1):92-103. doi: 10.1002/mds.29238. Epub 2022 Oct 14. PMID 36239376